CLINICAL TRIAL: NCT00442065
Title: A Study to Assess the Acute Technical Success of Aorfix™ Stent Grafts in the Treatment of Abdominal Aortic and Aorto-Iliac Aneurysm Where a Significant Degree of Vessel Angulation Exists at the Neck of the Aneurysm
Brief Title: ARBITER-II: Aorfix™ Bifurcated Safety and Performance Trial: Phase II, Angulated Vessels
Acronym: ARBITER-II
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lombard Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-001P2
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal aortic aneurysm study
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label, single arm (Active Comparator): A prospective, open label, single-arm (non-randomized) multi-center, international clinical device investigation to collect safety and performance data concerning the Aorfix™ Stent Graft System in the treatment of abdominal aortic aneurysm and aorto-iliac aneurysm where a significant degree of vessel angulation exists
  Interventions: Device: Aorfix™ Stent Grafts (AAA endovascular procedure)

INTERVENTIONS:
Device: Aorfix™ Stent Grafts (AAA endovascular procedure) — Endovascular treatment of AAA using the Aorfix™ Stent Graft and Delivery System
  Other Names: Aorfix™

SUMMARY:
To assess the safety and performance of Aorfix™ Stent Grafts in the treatment of Abdominal Aortic and Aorto-Iliac Aneurysm where a significant degree of vessel angulation exists at the neck of the aneurysm or in the common iliac arteries.

DETAILED DESCRIPTION:
The Aorfix™ Stent Graft is currently a CE-marked product indicated for AAA where the angle of the aneurysm is <65o. The objective of this study is to evaluate the safety and performance of the bifurcated Aorfix™ Stent Graft in the treatment of infrarenal abdominal aortic aneurysms and aorto-iliac aneurysms, in infrarenal necks angulated > 60o (between 60 to 90 degrees) as measured by 3-dimensional reconstruction in order to widen the indication.

The investigation is a prospective open label, single arm, multi-centre clinical study. The study group will consist of 25 evaluable participants. In order to account for patients lost to follow up (estimated at approximately 20%) up to 30 patients will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of abdominal aortic aneurysm 50 mm or larger in diameter, 40 mm or larger in diameter if symptomatic (i.e. pain, embolisation), or documented AAA growth of more than 5 mm within the previous 6 months, and/or including extension into common iliac artery(ies), or any saccular aneurysm.
* Infrarenal neck with a minimum length of 15 mm and a neck angulation between 60° and 90°, as assessed in 3 dimensions.
* The iliac artery diameter must be of appropriate diameter (1 mm smaller than the device diameter), with an appropriate distal landing length. The tortuosity of the common or external iliac arteries or femoral arteries must be low to medium (refer to operations manual).
* Patient provides written informed consent.
* Patients >18 years who are suitable for endovascular repair.
* Patient fit for endovascular surgery, with a diameter at the access sites of 7mm or larger bilaterally.
* Patient has a life expectancy longer than the duration of the study.

Exclusion Criteria:

* Patient has a ruptured aneurysm.
* Patient has insufficient length of proximal aneurysm neck (<15mm from aneurysm to lowest renal artery and <20 mm from the aneurysm to the SMA).
* Aneurysm extends above renal arteries.
* Proximal neck of aneurysm has significant loose thrombus associated with it, or significant circumferential calcifications.
* Pregnant or nursing patients.
* Patient unfit for bail-out surgery and appropriate anaesthesia.
* Patient with an acute or chronic aortic dissection or mycotic aneurysm (defined by localised asymmetric aneurysm sac).
* Patient has current non-localised infection.
* Patient has known allergy to graft materials, Nitinol, or contrast media.
* Patient's where imaging is problematic; an example is an obese patient.
* Patient has co-morbidities that deny vascular access, including small / tortuous access vessels.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoints are acute technical success, initial performance and safety at 1-month follow up. | 1-month post-procedure

SECONDARY OUTCOMES:
Secondary endpoints will examine recovery factors: operative time, ICU duration, blood loss, days to normal diet, days to discharge, days to ambulation, freedom from non-clinical events, need for secondary procedure and conversion to uni-iliac. | 6-months post-procedure
As well as safety at 6-month follow-up as measured by serious adverse events that occur up to 6-months post-procedure. | 6-months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: William C Loan, MD, FRCR, Principal Investigator — Belfast City Hospital Trust, Belfast, Ireland
Locations (6):
- 2 Interni Klinika; General University Hospital, Prague, Czechia
- Klinik für Gefäßchirurgie; St.-Franziskus Hospital Münster, Münster, Germany
- Department of Interventional Radiology, University School of Medicine, Lublin, Poland
- Vascular Surgery Division, Thoracic Institute, Hospital Clinic, University of Barcelona, Barcelona, Spain
- United Kingdom (2):
  - Belfast City Hospital Trust, Belfast
  - Freeman Hospital; Main X-Ray, Newcastle upon Tyne

REFERENCES:
- [Background] Harris PL, Vallabhaneni SR, Desgranges P, Becquemin JP, van Marrewijk C, Laheij RJ. Incidence and risk factors of late rupture, conversion, and death after endovascular repair of infrarenal aortic aneurysms: the EUROSTAR experience. European Collaborators on Stent/graft techniques for aortic aneurysm repair. J Vasc Surg. 2000 Oct;32(4):739-49. doi: 10.1067/mva.2000.109990. PMID 11013038